CLINICAL TRIAL: NCT01143233
Title: Suitability of an Infant Formula With Reduced Protein Content Based on a Partial Respectively an Extensive Proteinhydrolysate With and Without Pro- and Prebiotics for the Particular Nutritional Use by Infants.-Extension by 4 Year Follow-up
Brief Title: Low-protein Infant Formula With Partial or Extensive Proteinhydrolysate 4 Year Follow-up
Acronym: HippHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HiPP GmbH & Co. Vertrieb KG (Industry)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Hipp2010
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Disturbance of Growth

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- control formula group (Active Comparator): infants are fed a commercial, hydrolysed formula during the first 4 month of life, according to protocol
  Interventions: Other: control formula
- intervention formula 1 group (Experimental): infants are fed hydrolyzed infant formula with different protein content during the first 4 month of life, according to protocol
  Interventions: Other: intervention formula 1
- intervention formula 2 group (Experimental): infants are fed hydrolyzed infant formula with different protein content with pro- and prebiotics during the first 4 month of life, according to protocol
  Interventions: Other: intervention formula 2
- intervention formula 3 group (Experimental): infants are fed hydrolyzed instant formula with different protein content with pro- and prebiotics during the first 4 months of life, according to protocol
  Interventions: Other: intervention formula 3
- Reference group (No Intervention): infants are breast fed

INTERVENTIONS:
Other: control formula — infants are fed a commercial hydrolyzed formula
  Arms: control formula group
Other: intervention formula 1 — formula has hydrolysed protein and a different protein content
  Arms: intervention formula 1 group
Other: intervention formula 2 — formula has hydrolysed protein, different protein content and pro- and prebiotics
  Arms: intervention formula 2 group
Other: intervention formula 3 — formula has hydrolysed protein, different protein content and pro- and prebiotics
  Arms: intervention formula 3 group

SUMMARY:
The study is conducted to examine the suitability of partially respectively extensively hydrolyzed low protein infant formulae with and without pro- and prebiotics for healthy, term infants.

Primary hypothesis to be tested is: an infant formula based on a Protein hydrolysate with modified protein content is non inferior compared to a standard infant formula based on a Protein hyrolysate in respect to proper growth of healthy, term infants within the first four month of life.

4-year follow-up (without further Intervention) will focus on body composition and allergic predisposition.

DETAILED DESCRIPTION:
View Section Brief Summary

ELIGIBILITY:
Inclusion Criteria:

* written informed consent (by parents, caregiver)
* Healthy term newborns (gestational age: ≥ 37 weeks)
* Birth weight between 2.500 - 4.500 g
* Age at enrolment: < 28 days of age
* Infant received no other formula since birth
* Parents / Caregivers are able to speak German

Exclusion Criteria:

* Severe acquired or congenital illness
* preterm infants (gestational age < 37 weeks)
* Birth weight lower than 2.500 g or higher than 4.500 g
* Feeding a cows milk based formula or any other formula prior to inclusion in this study
* Participation in any other clinical study intervention
* Regular intake of supplementary pre- and probiotics by the child and/or breastfeeding mother
* Mothers with diabetes mellitus or mothers suffered from gestational diabetes
* Founded assumption that it will not be possible for parents / caregivers to be compliant with the study protocol
* Breastfed infants: illness of the mother, that may have an influence on the gastrointestinal tract of the child
* Breastfed infants: mother receives or received antibiotics one week before inclusion in this study or during the first study phase

Ages: 1 Day to 27 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 503 (Actual)
Dates: Start 2010-04; Primary Completion 2014-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
average weight gain | 4 months
  The intervention is to assess average weight gain in the first 4 months of life.

SECONDARY OUTCOMES:
allergic sensitization and symptoms | 12 months
  blood sample to assess allergic predisposition
Anthropometric data at age of 4 years | 4 years
  Weight, length and Head circumference measurements at Age of 4 years
Body composition (Skin fold) at age of 4 years | 4 years
  Caliper measurement at Age of 4 years
Body composition (fat mass, lean body mass) at age of 4 years | 4 years
  bioelectrical impedance Analysis at Age of 4 years
Allergic predisposition at age of 4 years by measuring specific IgE in blood | 4 years
  blood sample to allergic predisposition at Age of 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Wahn, Prof., Principal Investigator — Charité - Universitätsmedizin. Campus Virchow-Klinikum. Klinik für Pädiatrie mit Schwerpunkt Pneumologie/Immunologie; Kirsten Beyer, Prof, Principal Investigator — Charité - Universitätsmedizin. Campus Virchow-Klinikum. Klinik für Pädiatrie mit Schwerpunkt Pneumologie/Immunologie
Locations (5):
- Universitätsklinik für Kinder- und Jugendheilkunde, Abt. Neonatologie, päd. Intensivmedizin und Neuropädiatrie, Vienna, Austria
- Germany (3):
  - University Hospital Rostock, Rostock, Mecklenburg-Vorpommern
  - Klinik für Kinder- und Jugendmedizin der Ruhr-Universität Bochum, Bochum, North Rhine-Westphalia
  - Charité - Universitätsmedizin. Campus Virchow-Klinikum. Klinik für Pädiatrie mit Schwerpunkt Pneumologie/Immunologie, Berlin
- KBC "Dr Dragiša Mišović Dedinje", Belgrade, Serbia

REFERENCES:
- [Derived] Ahrens B, Hellmuth C, Haiden N, Olbertz D, Hamelmann E, Vusurovic M, Fleddermann M, Roehle R, Knoll A, Koletzko B, Wahn U, Beyer K. Hydrolyzed Formula With Reduced Protein Content Supports Adequate Growth: A Randomized Controlled Noninferiority Trial. J Pediatr Gastroenterol Nutr. 2018 May;66(5):822-830. doi: 10.1097/MPG.0000000000001853. PMID 29216020